CLINICAL TRIAL: NCT05613218
Title: Restrictive Versus Liberal Oxygenation Targets in Patients With Acute Heart Failure and Pulmonary Congestion - a Randomized Clinical Pilot-trial
Brief Title: Oxygen Targets in Acute Heart Failure With Pulmonary Congestion
Acronym: REDOX-AHF
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Johannes Grand, Principal Investigator, Copenhagen University Hospital, Hvidovre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REDOX
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Acute Heart Failure; Pulmonary Congestion; Hypoxemia
Keywords: acute heart failure; Pulmonary edema; Oxygen; Pulmonary congestion
MeSH Terms: conditions — Hypoxia; Pulmonary Edema | interventions — Oxygen

STUDY DESIGN:
Intervention Model Description: 1:1 allocation
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Oxygen-delivery will be given through a robot, which adjusts oxygen-flow towards a given oxygen-saturation target. The robots monitor will be turned of during the intervention and will only alarm in case of clinically relevant hypoxemia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liberal oxygenation group (Active Comparator): SpO2 target of 96%
  Interventions: Drug: Oxygen
- Restrictive oxygenation group (Active Comparator): SpO2 target of 90%.
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen — Patients will have nasal cannula or oxygen mask placed as the usual standard of care.
  Patients will be screened and randomized in the emergency department to either liberal or restrictive oxygenation after providing informed written consent and oxygen is titrated to the prespecified target range using an automated feedback device (O2MATIC). Consented patients will be randomly allocated to study groups via the web-based system within REDCap. The allocation will be concealed. Time at randomization will be considered as study time zero (T0). All patients will receive usual standard of care except for their O2 management. The intervention will last for 24 h. After 24 h, patients will be switched over to usual care for oxygen therapy. If the treating physician thinks, that the patient need another oxygenation target and it is thought to be harmful to continue with the allocated target, the intervention-phase can be stopped prematurely.

SUMMARY:
This investigator-initiated, prospective, randomized, blinded, multi-center, controlled trial will investigate the effect of a restrictive vs. liberal oxygenation-strategy in patients hospitalized with acute heart failure with pulmonary congestion.

Patients will be randomized 1:1 in the emergency department to either liberal or restrictive oxygenation after providing informed written consent.

1. Liberal oxygenation group = SpO2 target of 96%.
2. Restrictive oxygenation group = SpO2 target of 90%.

The allocation will be concealed through the use of an oxygen-delivery robot, termed O2MATIC. The study will include 122 patients.

DETAILED DESCRIPTION:
Background:

One million hospitalizations occur each year with a primary diagnosis of acute heart failure in the USA, with comparable numbers in Europe. Most patients with acute heart failure are treated with supplemental oxygen during hospitalization and guidelines recommend initiation of oxygen therapy if SpO2 <90% (class I, level C). However, no clinical trials of oxygen targets in humans with acute heart failure investigating clinically relevant endpoints have been performed.

Primary objective:

To investigate the effect of a restrictive vs. liberal oxygenation-strategy in patients hospitalized with acute heart failure.

Hypothesis:

Restrictive oxygenation is associated with improved clinical outcome compared to liberal oxygenation.

Design: Investigator-initiated, prospective, randomized, blinded, multi-center, controlled trial.

Intervention:

Patients will be randomized 1:1 in the emergency department to either liberal or restrictive oxygenation after providing informed written consent.

1. Liberal oxygenation group = SpO2 target of 96%.
2. Restrictive oxygenation group = SpO2 target of 90%.

Patients will have nasal cannula or oxygen mask placed as the usual care, and oxygen is titrated to the prespecified target range.

Consented patients will be randomly allocated to study groups via the automated web-based system within REDCap. The allocation will be concealed. Time at randomization will be considered as study time zero (T0). All patients will receive usual standard of care except for their oxygen-administration.

The intervention-phase will be 24 h, and hereafter oxygen therapy will be at the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Acute (within minutes to days) onset or worsening of subjective dyspnea
3. Oxygen saturation <92% (on arterial blood gas) or need of oxygen
4. At least one of the following clinical or radiological signs of congestion:

1. Pulmonary rales 2. Chest X-ray or CT with pulmonary congestion 3. Lung ultrasound with multiple B-lines

Exclusion Criteria:

1. More than 4 hours from hospital admission to randomization
2. Suspected infection or sepsis
3. Known severe pulmonary disease
4. Systolic blood pressure <90 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Pulmonary parenchymal fluid content after 24 hours | 24 hours
  Pulmonary parenchymal fluid content after 24 hours preceded by 10 minutes without oxygen-supplementation assessed noninvasively by the remote dielectric sensing (ReDS) device (Sensible Medical, Netanya, Israel)

SECONDARY OUTCOMES:
All-cause mortality | 30 days
  Death from all causes
Days alive out-of-hospital | 30 days
Time to freedom from oxygen-supplementation | 48 hours
4) Change from baseline in log-transformed biomarkers N-Terminal Pro-Brain Natriuretic Peptide to 24 hours from admission. | 24 hours
5) Arterial blood gas concentration after 24 hours preceded by 10 minutes without oxygen-supplementation. | 24 hours
Tricuspid annular plane systolic excursion | 24 hours
Global longitudinal strain of the right ventricle | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jens Hove, MD, PhD, Study Chair — Copenhagen University Hospital Amager-Hvidovre Department of Cardiology; Johannes Grand, MD, PhD, Principal Investigator — Copenhagen University Hospital Amager-Hvidovre Department of Cardiology; Ida Taraldsen, MD, Study Director — Copenhagen University Hospital Amager-Hvidovre Department of Cardiology
Locations (2):
- Denmark (2):
  - Bispebjerg Hospital, Copenhagen
  - Amager-Hvidovre Hospital, Copenhagen

IPD SHARING:
Plan to Share IPD: No